CLINICAL TRIAL: NCT04013529
Title: Connected Health to Decrease Opioid Use in Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01758
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participate in technology-enabled care without regret lottery
  Interventions: Behavioral: Way to Health technology enhanced care
- Experimental (Experimental): Participate in technology-enabled care with regret lottery
  Interventions: Behavioral: Regret lottery; Behavioral: Way to Health technology enhanced care

INTERVENTIONS:
Behavioral: Regret lottery — Subjects who achieve step goals are entered into a lottery in which they can win a financial incentive of $30 or $100.
  Arms: Experimental
Behavioral: Way to Health technology enhanced care — Subjects receive text reminders to reach activity goals.

SUMMARY:
The objective of this pilot study to evaluate if behavioral incentives applied at the VA Medical Center can appreciably increase participation in activities that promote mobility, and subsequently reduce pain severity and opioid use.

DETAILED DESCRIPTION:
Chronic pain is a highly prevalent and costly condition in the US. An estimated 88.5 million adults suffer from daily pain, resulting in estimated cost of $500- 635 biJlion due to lost productivity, and $261-300 billion in health care expenditures. To manage their chronic pain, 5 to 8 million Americans take an opioid medication daily. Yet , the risks associated with ongoing opioid prescription , including overdose, abuse and diversion, temper their analgesic effects.

Opioids are not more effective in the treatment of chronic pain compared with non-opioid approaches. Current guidelines have adapted to the evidence, recommending opioid-sparing approaches for treating patients with chronic pain, and tapering for those on higher doses to safer levels of use. Tapering opioids, however, requires replacing them with effective non-opioid strategies. Improving mobility has been shown to improve pain and decrease medication use among patients chronically prescribed opiates. Concurrently, financial incentives and the use of behavioral incentives have been shown to promote mobility.

Appreciating the gains in health outcomes that can be made with "connected health" approaches, we propose a novel pilot study designed to evaluate if technology enabled care (TEC) strategies and financial incentives can improve patient mobility in our chronic pain population, reduce pain and decrease opioid use . Our primary aim is to determine if chronic pain patients who receive TEC-enhanced treatment with financial incentives demonstrate increased participation in activities that promote mobility (physical therapy, yoga, tai chi) in comparison to patients receiving usual care. Secondary outcomes will include whether increased activity participation also reduces pain severity and opioid use, and improves function and increases the number of daily steps taken. The results of this pilot will enable us to determine what strategies are effective at increasing mobility and if these gains translate into reduced pain and decreased opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-malignant pain
* High dose opioid therapy
* Possession of activated cell phone with text messaging capabilities
* Willingness to comply with study requirements

Exclusion Criteria:

* Pain of malignant origin
* Sensory impairments precluding use of text messaging and activity tracker
* Physical disability precluding improvements in physical activity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Corporal Michael Cresenz VA Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Derived] Compton P, Chaiyachati KH, Dicks T, Medvedeva E, Chhabra M. A randomized controlled trial to evaluate a behavioral economic strategy for improving mobility in veterans with chronic pain. PLoS One. 2021 Oct 11;16(10):e0257320. doi: 10.1371/journal.pone.0257320. eCollection 2021. PMID 34634064

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Experimental
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.0) | 59.6 (13.5) | 57.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Activity Participation
Description: Stanford Exercise Questionnaire; min score = 0, max score = 180; higher scores = better outcome
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 19 | 19
score on a scale | 156.0 (116.8) | 135.8 (123.0)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Superiority; p = 0.90, ANCOVA

2. Primary Outcome: Increased Mobility
Description: steps per day measured by wearable step tracker at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Control | Experimental
Number analyzed (Participants) | 19 | 19
steps per day | 4313 (4231) | 4075 (5598)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Superiority; p = 0.88, ANCOVA

3. Secondary Outcome: Daily Opioid Use
Description: measured by opioid morphine mg equivalents used each day (MED)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: morphine mg equivalents per day (MED)
Arm/Group | Control | Experimental
Number analyzed (Participants) | 19 | 19
morphine mg equivalents per day (MED) | 167.2 (244.4) | 31.9 (35.53)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Superiority; p < 0.17, ANCOVA

4. Secondary Outcome: Physical Function
Description: measured by interference with walking on PROMIS (Patient-reported Outcomes Measurement Information System) pain interference tool, which is a 6-item self-report survey; each item is scored from 1 (not at all) to 5 (very much), thus scores ranged from 6 to 30, with higher score indicating more pain interference.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 19 | 19
units on a scale | 25.4 (10.94) | 24.2 (12.49)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Superiority; p < 0.05, ANCOVA

5. Secondary Outcome: Pain Severity
Description: measured by pain severity on PROMIS (Patient-reported Outcomes Measurement Information System) pain severity tool, which is a 3-item self-report survey; each item is scored from 1 (no pain at all) to 5 (very severity), thus scores ranged from 3 to 15, with higher score indicating more severe pain.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 19 | 19
units on a scale | 6.7 (1.63) | 6.8 (1.95)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Superiority; p = 0.81, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Although considered a minimal risk study, all participants were monitored for adverse events on a weekly basis.
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
Although subjects were blinded to group assignment, it is possible that those in the intervention arm communicated their potential to receive payment to those in the control arm who did not have the same benefit, which may have served as a disincentive for controls to engage in physical activity. Also, subjects in both groups received large numbers of text messages over the study period and may have found the messaging burdensome and thus stopped reading or responding to them as anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04013529/Prot_SAP_000.pdf